CLINICAL TRIAL: NCT04862585
Title: Safely Stopping Pre-Medications in Patients Receiving Paclitaxel: A Randomized Trial
Brief Title: Safely Stopping Pre-medications in Patients With Breast Cancer Who Are Receiving Paclitaxel
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Michael Berger, PharmD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-20429; NCI-2021-01586 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Breast Carcinoma; Prognostic Stage 0 Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms | interventions — Cimetidine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Diphenhydramine; Famotidine; Paclitaxel; Taxes; Ranitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (paclitaxel, pre-medications) (Active Comparator): Patients continue on pre-medications (dexamethasone, diphenhydramine, famotidine/ranitidine/cimetidine) with all future doses of paclitaxel.
  Interventions: Drug: Cimetidine; Drug: Dexamethasone; Drug: Diphenhydramine; Drug: Famotidine; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Drug: Ranitidine
- Arm II (paclitaxel) (Experimental): Patients discontinue premedications (dexamethasone, diphenhydramine, famotidine/ranitidine/cimetidine) with all future doses of paclitaxel, unless patient develops a subsequent infusion HSR.
  Interventions: Drug: Paclitaxel; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Cimetidine — Given IV and/or PO
  Other Names: Tagamet
  Arms: Arm I (paclitaxel, pre-medications)
Drug: Dexamethasone — Given IV and/or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Arm I (paclitaxel, pre-medications)
Drug: Diphenhydramine — Given IV and/or PO
  Other Names: FAR 90X2; PM 255; Probedryl; Rigidyl; S51; Syntedril
  Arms: Arm I (paclitaxel, pre-medications)
Drug: Famotidine — Given IV and/or PO
  Other Names: Pepcid; Pepcid AC
  Arms: Arm I (paclitaxel, pre-medications)
Drug: Paclitaxel — Weekly or every 14 day dosing
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Ranitidine — Given IV and/or PO
  Arms: Arm I (paclitaxel, pre-medications)

SUMMARY:
This phase II/III trial investigates the difference in rates of infusion hypersensitivity reaction in patients with breast cancer who are receiving paclitaxel alone or in combination with other cancer drugs which require parenteral rescue medication after stopping standard pre-medications (dexamethasone, diphenhydramine, famotidine/cimetidine/ranitidine), compared to continuing premedications. Paclitaxel is a drug used to treat breast cancer, ovarian cancer, and autoimmune deficiency syndrome (AIDS)-related Kaposi sarcoma. It blocks cell growth by stopping cell division and may kill cancer cells. It is a type of antimitotic agent. However, there are side-effects and toxicities associated with repeat exposure to this pre-medication regimen. With prolonged use of paclitaxel, especially during weekly regimens, patients are exposed to repeat doses of drugs that prevent hypersensitivity reactions. Side effects include, but are not limited to, insomnia, gastritis, fluid retention, weight gain, mood changes and immune suppression. The information gained from this study may positively influence clinical practice and help researchers develop methods to safely stop pre-medications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the difference in rates of infusion hypersensitivity reaction (HSR) requiring parenteral rescue medications following the discontinuation of pre-medications after 2 doses of paclitaxel, compared to continuing premedications, in breast cancer patients who have not experienced an infusion HSR with their first 2 paclitaxel doses.

OUTLINE:

Patients receive paclitaxel per standard of care as a single agent or in combination with dexamethasone intravenously (IV) and/or orally (PO), diphenhydramine IV and/or PO and either famotidine IV and/or PO, ranitidine IV and/or PO or cimetidine IV and/or PO. Patients who don't experience any infusion hypersensitivity reaction after the first 2 doses of paclitaxel are randomized to 1 of 2 arms.

ARM I (STANDARD OF CARE): Patients continue on pre-medications (dexamethasone, diphenhydramine, famotidine/ranitidine/cimetidine) with all future doses of paclitaxel.

ARM II (EXPERIMENTAL): Patients discontinue premedications (dexamethasone, diphenhydramine, famotidine/ranitidine/cimetidine) with all future doses of paclitaxel, unless patient develops a subsequent infusion HSR.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to receive at least 4 doses of paclitaxel as a single-agent or in combination with trastuzumab, pertuzumab, bevacizumab, pembrolizumab, lapatinib, gemcitabine or other drug combination (excluding cisplatin or carboplatin) for the treatment of any stage, histologically confirmed breast cancer
* Ability to complete questionnaires by themselves or with assistance
* Life expectancy > 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Age >= 18
* Able to give informed consent
* Patients must be scheduled to receive prophylactic HSR premedications (IV or oral) consisting of a histamine-1 (H1) antagonist (diphenhydramine) or cetirizine (a histamine-1 (H1) antagonists), dexamethasone (a steroid) and a either famotidine, ranitidine or cimetidine (histamine-2 (H2) antagonists), per institutional guidelines, prior to each of their first 2 doses of paclitaxel
* Patients may enroll, or currently be enrolled in another concurrent clinical trial provided the other trial would not prohibit the discontinuation of paclitaxel premedications

Exclusion Criteria:

* Patients who have received at least 1 prior lifetime dose of paclitaxel or paclitaxel albumin-bound
* Patients receiving paclitaxel in combination with carboplatin or cisplatin (due to risk of hypersensitivity with platinum compounds)
* History of grade 3 hypersensitivity reaction to Cremophor EL containing medications (e.g. paclitaxel, cyclosporine, ixabepilone, teniposide)
* Patients receiving therapeutic daily doses of systemic corticosteroids. Intermittent oral steroids for nausea or for acute inflammatory conditions (i.e. methylprednisolone dosepak) and inhaled, intranasal or topical corticosteroids are permitted
* Patients who are pregnant or nursing. Paclitaxel is classified by the Food and Drug Administration (FDA) as "pregnancy category D". Pregnancy testing (urine or blood human chorionic gonadotropin [Hcg]) will be done and documented prior to enrollment if pregnancy is clinically suspected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Berger, Pharm.D., Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 130 subjects enrolled. 32 not randomized (29 experienced HSR in 1st or 2nd dose of Taxol, 1 ineligible, 2 withdrew). 98 randomized: 50 randomized to continue premeds (4 withdrew after randomization) total of 46 evaluable. 48 randomized to stop premeds (5 withdrew after randomization) total of 43 evaluable.
Period: Overall Study
Arm/Group | Arm I (Paclitaxel, Pre-medications) | Arm II (Paclitaxel)
Started | 50 | 48
Completed | 46 | 43
Not Completed | 4 | 5
Not completed — two subjects withdrew due to perceived side effects of premedications | 2 | 0
Not completed — five subjects withdrew due to what they considered to be an unfavorable randomization assignment | 2 | 3
Not completed — one subject discontinued paclitaxel due to toxicity | 0 | 1
Not completed — one withdrew without providing a reason | 0 | 1

BASELINE CHARACTERISTICS:
Population: 130 subjects enrolled. 32 not randomized (29 experienced HSR in 1st or 2nd dose of Taxol, 1 ineligible, 2 withdrew). 98 randomized: 50 randomized to continue premeds (4 withdrew after randomization) total of 46 evaluable. 48 randomized to stop premeds (5 withdrew after randomization) total of 43 evaluable.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Paclitaxel, Pre-medications) | Arm II (Paclitaxel) | Total
Number analyzed (Participants) | 46 | 43 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 34 | 69
  >=65 years | 11 | 9 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 43 | 88
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 46 | 42 | 88
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 7 | 8
  White | 45 | 33 | 78
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 46 | 43 | 89

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Grade 2 or Greater Reactions That Require Parenteral Rescue Medications to Treat an Infusion Hypersensitivity Reaction (HSR) After the First 2 Doses of Paclitaxel With or Without Continued Premedication Dosing
Description: The proportion of patients having infusion HSR of grade 2 or greater requiring parental treatment (rescue medications) will be estimated along with a 95% confidence interval. The difference in proportions of patients with grade 2 or greater infusion HSR needing rescue medication will be estimated along with a 95% confidence interval using the Z-test of normal approximations of the binomial distributions. As a sensitivity analysis, will repeat the analysis including patients assigned to the discontinuation arm but decided to restart pre-medications and patients assigned to the continuation arm but demanded to have premedications discontinued as having experienced HSR.
Time Frame: Up to 2 years and 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Paclitaxel, Pre-medications) | Arm II (Paclitaxel)
Number analyzed (Participants) | 46 | 43
Participants | 0 | 1

2. Secondary Outcome: Correlation Between Abbreviated Premedication Regimen Results to Quality of Life (QoL)
Description: Will determine whether an abbreviated pre-medication regimen results in an improvement in patient-reported quality of life, as measured by an 11-point numerical analog scale (scores range from 0-10 with higher values representing a worse QoL). Both "undesirable appetite increase" and "reported rash" will be rated on this 11-point scale from 0 to 10 with higher values representing a worse undesirable appetite or a worse rash. The "worst reported undesirable appetite increase" and "worst reported rash" scores representing the highest mean score reported at an individual time point for each arm, will be summarized. In addition the change from baseline will be summarized by mean separately by treatment arm. Data will be captured every day, for one week after each dose of chemotherapy.
Time Frame: Up to 2 years and 8 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm I (Paclitaxel, Pre-medications) | Arm II (Paclitaxel)
Number analyzed (Participants) | 46 | 43
score on a scale
  Worst reported undesirable appetite increase | 2.5 [1.77 to 3.23] | 1 [0.54 to 1.46]
  Worst reported rash | 3.3 [2.58 to 4.12] | 2.3 [1.48 to 3.13]
  Change in undesirable appetite increase from baseline | 1.7 [1.08 to 2.36] | 0.5 [0.15 to 0.80]
  Change in reported rash from baseline | 2.9 [2.11 to 3.72] | 1.9 [1.13 to 2.59]

3. Other Pre Specified Outcome: Differences in a Number of Symptoms That Might be Improved, or Worsened, by the Hypersensitivity Prevention Drugs
Description: Each symptom will be summarized by median (range) at each time point by treatment arm and the weekly average will be compared between arms using the Wilcoxon rank sum test.
Time Frame: Up to 6 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: The Number of Patients Who, After Discontinuing Pre-medications, Request That the Premedications be Resumed to Ameliorate Side-effects That the Patient Thinks Have Worsened Since Premedications Were Stopped (i.e. Nausea, Rash, Arthralgia)
Description: The frequency and percentages of patients who, after discontinuing pre-medications, request that the pre-medications be resumed to ameliorate side-effects that the patient thinks have worsened since pre-medications were stopped (i.e. nausea, rash, arthralgia) will be summarized.
Time Frame: Up to 6 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Weight Changes Across Study Periods for Both Arms of the Study
Description: Weight changes over time will be summarized at each time point using mean (standard deviation) and plotted by treatment arm. Weight change from baseline to 10 weeks post-randomization will be compared between arms that receive weekly paclitaxel using a t-test of two independent samples.
Time Frame: Up to 6 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: The Impact of Patient Self-reported Allergies
Description: Will report the impact of patient self-reported allergies, prior to starting paclitaxel (2 or more versus 3 or less), on the incidence of infusion HSR and rescue medication usage. Frequency of patient self-reported allergies (2 or more versus less) on the incidence of infusion HSR and rescue medication usage will be tabulated.
Time Frame: Up to 6 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Patient Outcomes
Description: The rates of rescue medication by arms will be estimated by race/ethnicity group to explore whether there is a differential effect from stopping hypersensitivity reaction by race/ethnicity.
Time Frame: Up to 6 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: adverse events not collected for this study
Description: adverse events not collected for this study
Arm/Group | Arm I (Paclitaxel, Pre-medications) | Arm II (Paclitaxel)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT04862585/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT04862585/ICF_001.pdf